CLINICAL TRIAL: NCT06881225
Title: Study on the Regulation of Blood-Brain Barrier Permeability by APOE Gene Polymorphism and Its Impact on Cognitive Function After Radiotherapy for Nasopharyngeal Carcinoma: an MRI Investigation
Brief Title: Regulation of Blood-Brain Barrier Permeability by APOE Gene Polymorphism and Its Impact on Cognitive Function Post-Radiotherapy in Nasopharyngeal Carcinoma: an MRI Study
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaofei Lv, President, Sun Yat-sen University
Other Study IDs: G2024-069-01
Record Dates: First submitted 2025-02-15; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Using DCE-MRI, fMRI, and DSI, establish a longitudinal brain functional and structural imaging database for three groups of nasopharyngeal carcinoma patients before and 18 months after radiotherapy. — 1. Resting-state fMRI:
     Use the Gradient Echo Echo Planar Imaging (GRE-EPI) sequence with the following parameters: repetition time (TR) = 2000 ms, echo time (TE) = 30 ms, flip angle (FA) = 90°, slice thickness = 3.0 mm, slice spacing = 0.8 mm, field of view (FOV) = 240 mm × 240 mm, matrix = 128 × 128, in-plane resolution = 64 × 64, 39 axial slices scanned, 240 dynamic scans.
  2. DSI:
     Use diffusion-sensitive imaging (DSI) with 64 diffusion directions, b-values of 0 and 1000 s/mm², TR = 3000 ms, TE = 64 ms, number of excitations (NEX) = 1, matrix = 112 × 112, FOV = 224 mm × 224 mm, slice thickness = 2 mm, no spacing between slices, full brain coverage, and 75 slices scanned.
  3. Three-dimensional brain structural MRI:
  Sagittal data acquisition is performed with the following parameters: TR = 8.16 ms, TE = 3.18 ms, inversion time (TI) = 800 ms, flip angle (FA) = 8°, matrix = 256 × 256, FOV = 256 mm × 256 mm, voxel size = 1 mm × 1 mm × 1 mm, and 176 slices scanned.

SUMMARY:
adiotherapy-induced cognitive dysfunction is a severe complication following radiotherapy for nasopharyngeal carcinoma (NPC). Our previous studies have demonstrated that abnormalities in brain function and structural connectivity after radiotherapy play a significant role in the occurrence of radiation-induced cognitive dysfunction. However, the key risk factors and underlying neural mechanisms remain unclear. Research has shown that increased blood-brain barrier (BBB) permeability after radiotherapy is an important mechanism leading to cognitive dysfunction, and different APOE gene subtypes can regulate BBB permeability. Therefore, APOE gene polymorphisms are likely to influence post-radiotherapy vascular barrier permeability in NPC patients, thereby affecting their brain function and structural connectivity changes, and ultimately impacting their cognitive function.

This project aims to establish a longitudinal brain imaging database for NPC patients with different APOE genotypes before and after radiotherapy, based on previous research findings. The project will integrate dynamic contrast-enhanced MRI (DCE-MR), resting-state functional MRI (fMRI), and diffusion spectrum imaging (DSI) techniques. By comparing DCE-derived metrics across different genotype groups, the study seeks to identify brain regions with BBB damage differences between APOE genotype groups before and after radiotherapy. Furthermore, it will investigate how BBB damage in these brain regions mediates functional and structural connectivity abnormalities, and their relationship with radiation-induced cognitive dysfunction. The goal is to clarify the neural regulation mechanism of APOE gene polymorphisms in radiation-induced cognitive dysfunction and to identify risk factors for radiation-induced cognitive dysfunction. This research will provide a theoretical basis and valuable reference for the individualized prevention and treatment of radiation-induced cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Patients newly diagnosed with nasopharyngeal carcinoma, pathologically confirmed, and who have not received anti - tumor treatments such as surgery, induction chemotherapy, or radiotherapy.

All patients are of Han ethnicity and right - handed. Patients are aged between 20 and 60 years old, with an educational level of junior high school or above.

The clinical stage of the included patients is AJCC 8th edition stage I - IVa, without distant metastasis, and patients are scheduled to receive intensity - modulated radiotherapy (IMRT) according to the clinical plan.

Patients have no other serious systemic diseases except nasopharyngeal carcinoma.

There is no intracranial invasion of nasopharyngeal carcinoma. Routine MRI examinations (including T1WI, T2WI, and FLAIR) are negative. The baseline basic cognitive assessment scales (MoCA and MMSE) before radiotherapy are normal.

Patients have no family history of mental illness. Patients have no history of neurological diseases or head trauma. After fully understanding the experimental content, the subjects agree to participate in this project and sign the informed consent form

Exclusion Criteria:

Patients diagnosed with Alzheimer's disease (AD) before being included. AD is diagnosed by psychiatrists according to the 9th Revision of the International Classification of Diseases, Clinical Modification (ICD - 9 - CM).

Patients with intracranial lesions detected by routine MRI examinations. Patients with contraindications to magnetic resonance examinations. Patients with concurrent other diseases. Patients with tumor recurrence who need re - radiotherapy, or those who cannot adhere to and complete IMRT treatment.

Left - handed or ambidextrous patients. Patients with a history of head trauma or mental/neurological diseases. Patients aged less than 20 or more than 60 years old. Patients with serious systemic diseases such as heart, lung, or kidney diseases.

Patients with diabetes or hypertension. Patients who cannot cooperate to complete the neurocognitive scale tests.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Collect nasopharyngeal carcinoma patients who seek medical treatment at Sun Yat - sen University Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood-Brain Barrier Permeability as Measured by Ktrans Values from DCE-MRI | From enrollment to 18 months after the completion of radiotherapy
  The change in blood-brain barrier permeability will be quantified using the volume transfer constant (Ktrans) derived from Dynamic Contrast-Enhanced MRI (DCE-MRI). Ktrans values will be measured at baseline (pre-radiotherapy) and at 18 months post-radiotherapy. The difference in Ktrans values between these time points will be calculated to assess the change in permeability.
Change in Functional Connectivity as Measured by Resting-State fMRI | From enrollment to 18 months after the completion of radiotherapy
  Functional connectivity will be assessed using resting-state functional MRI (fMRI). The strength of functional connections between specific brain regions, particularly those identified as having significant blood-brain barrier damage, will be measured at baseline and at 18 months post-radiotherapy. The change in functional connectivity strength will be calculated and reported.
Change in Structural Connectivity as Measured by Diffusion Spectrum Imaging (DSI) | From enrollment to 18 months after the completion of radiotherapy
  Structural connectivity will be evaluated using Diffusion Spectrum Imaging (DSI). The integrity of white matter tracts, particularly those connecting regions with significant blood-brain barrier damage, will be measured at baseline and at 18 months post-radiotherapy. The change in structural connectivity, as indicated by metrics such as fractional anisotropy (FA) and mean diffusivity (MD), will be calculated and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Imaging, Sun Yat-sen University Cancer Center, State Key Laboratory of Oncology in South China, Collaborative Innovation Center for Cancer Medicine, Guangdong Key Laboratory of Nasopharyngeal Carcinoma Diagnosis and Therapy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lozupone M, Imbimbo BP, Balducci C, Lo Vecchio F, Bisceglia P, Latino RR, Leone M, Dibello V, Solfrizzi V, Greco A, Daniele A, Watling M, Seripa D, Panza F. Does the imbalance in the apolipoprotein E isoforms underlie the pathophysiological process of sporadic Alzheimer's disease? Alzheimers Dement. 2023 Jan;19(1):353-368. doi: 10.1002/alz.12728. Epub 2022 Jul 28. PMID 35900209
- [Background] Main BS, Villapol S, Sloley SS, Barton DJ, Parsadanian M, Agbaegbu C, Stefos K, McCann MS, Washington PM, Rodriguez OC, Burns MP. Apolipoprotein E4 impairs spontaneous blood brain barrier repair following traumatic brain injury. Mol Neurodegener. 2018 Apr 4;13(1):17. doi: 10.1186/s13024-018-0249-5. PMID 29618365
- [Background] Jackson RJ, Meltzer JC, Nguyen H, Commins C, Bennett RE, Hudry E, Hyman BT. APOE4 derived from astrocytes leads to blood-brain barrier impairment. Brain. 2022 Oct 21;145(10):3582-3593. doi: 10.1093/brain/awab478. PMID 34957486
- [Background] Bell RD, Winkler EA, Singh I, Sagare AP, Deane R, Wu Z, Holtzman DM, Betsholtz C, Armulik A, Sallstrom J, Berk BC, Zlokovic BV. Apolipoprotein E controls cerebrovascular integrity via cyclophilin A. Nature. 2012 May 16;485(7399):512-6. doi: 10.1038/nature11087. PMID 22622580
- [Background] Tang Y, Luo D, Rong X, Shi X, Peng Y. Psychological disorders, cognitive dysfunction and quality of life in nasopharyngeal carcinoma patients with radiation-induced brain injury. PLoS One. 2012;7(6):e36529. doi: 10.1371/journal.pone.0036529. Epub 2012 Jun 11. PMID 22701557
- [Background] Penn IW, Chung CH, Huang YC, Chen MC, Sun CA, Yip PK, Chien WC. Increased risk of dementia in patients with nasopharyngeal cancer treated with radiation therapy: A nationwide population-based cohort study. Arch Gerontol Geriatr. 2021 Mar-Apr;93:104303. doi: 10.1016/j.archger.2020.104303. Epub 2020 Nov 22. PMID 33302001
- [Background] McDowell LJ, Ringash J, Xu W, Chan B, Lu L, Waldron J, Rock K, So N, Huang SH, Giuliani M, Hope A, O'Sullivan B, Bratman SV, Cho J, Kim J, Jang R, Bayley A, Bernstein LJ. A cross sectional study in cognitive and neurobehavioral impairment in long-term nasopharyngeal cancer survivors treated with intensity-modulated radiotherapy. Radiother Oncol. 2019 Feb;131:179-185. doi: 10.1016/j.radonc.2018.09.012. Epub 2018 Sep 29. PMID 30279047
- [Background] Zheng Z, Wang B, Zhao Q, Zhang Y, Wei J, Meng L, Xin Y, Jiang X. Research progress on mechanism and imaging of temporal lobe injury induced by radiotherapy for head and neck cancer. Eur Radiol. 2022 Jan;32(1):319-330. doi: 10.1007/s00330-021-08164-6. Epub 2021 Jul 29. PMID 34327577
- [Background] Hsiao KY, Yeh SA, Chang CC, Tsai PC, Wu JM, Gau JS. Cognitive function before and after intensity-modulated radiation therapy in patients with nasopharyngeal carcinoma: a prospective study. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):722-6. doi: 10.1016/j.ijrobp.2009.06.080. Epub 2010 Jan 13. PMID 20044217
- [Background] Tofilon PJ, Fike JR. The radioresponse of the central nervous system: a dynamic process. Radiat Res. 2000 Apr;153(4):357-70. doi: 10.1667/0033-7587(2000)153[0357:trotcn]2.0.co;2. PMID 10798963